CLINICAL TRIAL: NCT02957500
Title: To Evaluate Anti-adhesive Effect and Safety of a Mixed Solid of Poloxamer, Gelatin and Chitosan(Mediclore®) After Intrauterine Surgery in Patient With Gynecological Disease, a Multicenter, Randomized, Double- Blinded Study
Brief Title: To Evaluate Anti-adhesive Effect and Safety of a Mixed Solid of Poloxamer, Gelatin and Chitosan(Mediclore®)
Acronym: antiadhesion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CGBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CG-AHS007
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2016-11

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mediclore® (Experimental): adhesion barrier Mediclore 5cc, to apply medical device fully around intrauterine surgery area
  Interventions: Device: Mediclore® (adhesion barrier)
- No treatment (No Intervention): standard treatment for surgery

INTERVENTIONS:
Device: Mediclore® (adhesion barrier)
  Arms: Mediclore®

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Mediclore®, as an antiadhesive barrier, which is made of Poloxamer, Gelatin and Chitosan.

DETAILED DESCRIPTION:
to evaluate the efficacy and safety of Mediclore®, as an antiadhesive barrier

ELIGIBILITY:
Inclusion Criteria:

* the patients with submucosal myomas, endometrial polyps, intra-uterine adhesion, uterine septa, dysfunctional uterine bleeding
* Written informed consent
* Patients without clinically significant lab

Exclusion Criteria:

* having enrolled another clinical trials within 1 month
* Immunosuppression or autoimmune disease
* Anticoagulant, general steroids within a week from surgery
* Incompatible medications
* Serious diseases (heart failure, renal failure, liver failure, uncontrolled hypertension, diabetes mellitus, coagulation deficiencies)

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2016-11-22 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Adhesion incidence rate following 4 weeks | 4weeks

CONTACTS AND LOCATIONS:
Locations (1):
- CHA kangnam medical center, CHA university, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
undecided